CLINICAL TRIAL: NCT03432247
Title: Mechanisms of Music Therapy to Palliate Pain in Patients With Advanced Cancer
Brief Title: Pain Management Support Study for Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Joke Bradt, Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01NR016681 (NIH); 1R01NR016681-01A1 (NIH)
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Advanced Cancer
Keywords: music therapy; bone pain; pain management; advanced cancer
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Music Therapy (Experimental): Six 45-minute individual interactive music therapy sessions.
  Interventions: Behavioral: Interactive Music Therapy
- Verbal-based support (Active Comparator): Six 45-minute individual verbal support sessions
  Interventions: Behavioral: Verbal support

INTERVENTIONS:
Behavioral: Interactive Music Therapy — Six 45-minute individual interactive music therapy (IMT) sessions delivered by a board-certified music therapist. Sessions start with music-guided breathing, imagery, or humming. The music therapist then engages the participant in singing of familiar songs and co-created vocal or instrumental music improvisations based on patient needs. Discussion about the meaning assigned to songs and emotions expressed through the improvisations follow. The IMT experiences are aimed at facilitating emotional expression, offering support through interactive music making, and strengthening inner resources of creativity. In addition, each week the participant learns music-based techniques for self-management of anxiety, stress, mood, and pain.
  Arms: Interactive Music Therapy
Behavioral: Verbal support — Six 45-minute individual sessions delivered by a master's level clinician with training in counseling. The sessions are focused on patient-initiated conversations about their pain, life stressors and the impact on their daily life. The intervener provides nondirective, supportive care by offering supportive, validating statements and reflective listening. The intervener refrains from employing active suggestion, problem-solving or behavioral or cognitive therapy techniques. The verbal support sessions are aimed at providing an empathic, therapeutic environment to facilitate emotional expression and sharing of worries and fears.
  Arms: Verbal-based support

SUMMARY:
Chronic pain is one of the most feared symptoms in people with cancer. Insufficient relief from pharmacological treatments and the fear of side effects are important reasons for the growing use of complementary pain management approaches in cancer care. On such approach is music therapy. Although several studies have demonstrated that music therapy interventions can reduce pain in people with cancer, few studies have examined the therapeutic mechanisms that explain how music therapy interventions lead to improved pain management. The purpose of this study is to examine whether an interactive music therapy intervention improves psychological and social factors that play an important role in chronic pain management in people with advanced cancer. The findings will contribute towards the optimization of music therapy for palliation of chronic pain in people with advanced cancer.

DETAILED DESCRIPTION:
This study addresses the public health problem of chronic pain as one of the most feared symptoms in people with cancer, with 70% to 90% of patients with advanced disease reporting pain. Unrelieved pain remains a challenge in cancer care. Insufficient relief from pharmacological treatments and the fear of side effects are important reasons for the growing use of complementary pain management approaches in people with cancer. One such approach is music therapy. Although efficacy of music therapy for pain has been established, there are no mechanistic studies clarifying how it works in clinical populations. Thus, there is a lack of knowledge related to 1) therapeutic mechanisms that lead to improvement (mediator effects) and 2) the relationship between patient characteristics and treatment response (moderator effects). Yet, it is well accepted that knowledge of mediators and moderators as well as a validated theory of action (i.e., how the intervention activates the mediators) are needed to optimize psychosocial treatment interventions. Therefore, the overarching goals of this study are to 1) examine mediators and moderators hypothesized to account for the pain-reducing effects of Interactive Music Therapy (IMT) in people with advanced cancer and chronic pain and 2) validate IMT's theory of action. The mediation model to be tested in this study aligns with a biopsychosocial framework to palliation of chronic pain and is based on findings from a preliminary study. The investigators postulate that anxiety, mood, self-efficacy and perceived support mediate the effects of IMT on pain outcomes (i.e. pain intensity and pain interference). In addition, the impact of several moderators on the hypothesized mediation model, namely adult playfulness, perceived musical competence, and treatment expectancy, will be tested. This study uses a mixed methods intervention design in which qualitative data (i.e. semi-structured follow-up interviews) are embedded within a randomized controlled trial. A total of 100 outpatients with advanced cancer and chronic bone pain will be randomized to one of two 6-week treatments: 1) Interactive Music Therapy or 2) Verbal-based support. The mediators and pain outcomes will be measured at baseline and after the fourth and sixth session using self-report measures as well as biomarkers (salivary cortisol, lachrymal dopamine content, serum oxytocin, and plasma β-endorphins). Follow-up interviews with a subsample of 30 participants will enable the investigators to examine the congruence between the hypothesized mediators and moderators and participant explanations of how IMT influences chronic pain management (i.e. theory of action). This study will contribute towards the optimization of music therapy for palliation of chronic pain in people with advanced cancer through a better understanding of the impact of mediators and moderators of IMT on chronic pain management. The results of this study will provide estimated effects sizes of IMT on the mediators and preliminary effect size estimates for the pain outcomes. This information will be instrumental in the development of a subsequent large-scale efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* male or female outpatients with advanced cancer (Stage 3 & 4; or relapse refractory patients for myeloma)
* diagnosed with locally advanced cancer that has extended to organs/soft tissue or is impinging on or eroding the bone; or bone metastases or soft tissue metastasis
* moderate to severe pain with an average intensity ≥4 on a 0-10 Numeric Rating Scale (NRS)
* experiencing pain for ≥ 3 months
* Karnofsky Performance score of ≥ 60 or the Eastern Cooperative Group Performance Status (ECOG) equivalent of ≤ 2 (i.e. requires occasional assistance, but is able to care for most of their personal needs)

Exclusion Criteria:

* expected survival ≤ 3 months
* primary central nervous system (CNS) tumor or CNS metastatic disease that impairs concentration, memory, balance or focus that would preclude ability to participate in a 60 minute, recurring activity and completion of self-report measures
* hematologic malignancies except for myeloma which causes significant bone pain
* ≤ 3 weeks post-operation from start of study
* active psychosis or dementia
* inability to speak or write English
* moderate to severe hearing impairment
* current smoking
* current alcohol dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | through study completion, a maximum of 12 weeks
  measured by PROMIS® Pain Intensity-Short Form (SF)3a
Pain Interference | through study completion, a maximum of 12 weeks
  measured by PROMIS® Cancer-Pain Interference -SF 6b
Patient Perception of Change | through study completion, a maximum of 12 weeks
  measured by Patient Global Impression of Change Scale (PGIC)
Serum β-endorphin | through study completion, a maximum of 12 weeks
  biomarker for pain intensity

SECONDARY OUTCOMES:
Anxiety | through study completion, a maximum of 12 weeks
  Mediator outcome measured by PROMIS® Cancer-Anxiety - SF
Mood | through study completion, a maximum of 12 weeks
  Mediator outcome measured by Positive and Negative Affect Scale (PANAS)
Perceived support | through study completion, a maximum of 12 weeks
  Mediator outcome measured by PROMIS® Emotional Support - SF 6a
Self-efficacy | through study completion, a maximum of 12 weeks
  Mediator outcome measured by PROMIS® Self-Efficacy of Symptoms
Salivary cortisol | through study completion, a maximum of 12 weeks
  Mediator outcome (biomarker for anxiety)
Serum oxytocin | through study completion, a maximum of 12 weeks
  Mediator outcome (biomarker for social support)
Lachrymal dopamine | through study completion, a maximum of 12 weeks
  Mediator outcome (biomarker for mood)

OTHER OUTCOMES:
Treatment expectancy | Baseline
  Moderator outcome measured by Credibility/Expectancy Questionnaire (CEQ)
Perceived Musical Competence | Baseline
  Moderator outcome measured by two-item questionnaire
Adult playfulness | Baseline
  Moderator outcome measured by Short Measure for Adult Playfulness (SMAP)

CONTACTS AND LOCATIONS:
Overall Officials: Joke Bradt, PhD, Principal Investigator — Drexel University
Locations (3):
- United States (3):
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Cancer Treatment Centers of America (CTCA), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We will make the de-identified datasets available to other researchers. Researchers will be asked to submit a formal request for data sharing to the PI that outlines the purpose of the secondary data analysis. Data and associated documentation will be made available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol
Time Frame: After completion of study report and publication of results
Access Criteria: We will make the de-identified datasets available to other researchers. Researchers will be asked to submit a formal request for data sharing to the PI that outlines the purpose of the secondary data analysis. Data and associated documentation will be made available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Bradt J, Leader A, Worster B, Myers-Coffman K, Bryl K, Biondo J, Schneible B, Cottone C, Selvan P, Zhang F. Music Therapy for Pain Management for People With Advanced Cancer: A Randomized Controlled Trial. Psychooncology. 2024 Oct;33(10):e70005. doi: 10.1002/pon.70005. PMID 39450934